CLINICAL TRIAL: NCT00177892
Title: OSA and Metabolic Syndrome: Role of Oxidative Stress
Brief Title: Obstructive Sleep Apnea (OSA) and Metabolic Syndrome: Role of Oxidative Stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Mark H Sanders, MD, University of Pittsburgh School of Medicine
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: AG0089; 5R01AG023977 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Obstructive Sleep Apnea; Metabolic Syndrome X
Keywords: Sleep fragmentation; Intermittent hypoxia; Obstructive Sleep Apnea; Metabolic Syndrome; Insulin resistance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Metabolic Syndrome; Sleep Deprivation; Insulin Resistance | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): non-OSAH/overweight individuals with the Metabolic Syndrome
  Interventions: Procedure: sleep disruption
- 2 (Experimental): non-OSAH/overweight individuals without Metabolic Syndrome
  Interventions: Procedure: sleep disruption
- 3 (Active Comparator): non-OSAH/normal weight without Metabolic Syndrome
  Interventions: Procedure: sleep disruption
- 4 (Experimental): OSAH patients with chronic positive airway pressure therapy
  Interventions: Procedure: sleep with and without positive pressure
- 5 (Experimental): OSAH patients without chronic positive airway pressure therapy
  Interventions: Procedure: sleep with and without positive pressure

INTERVENTIONS:
Procedure: sleep disruption — experimentally-induced Sleep Fragmentation
  Arms: 1; 2; 3
Procedure: sleep with and without positive pressure — OSAH patients with and without chronic positive airway pressure therapy
  Other Names: fragmentation + normoxia; fragmentation + hypoxia
  Arms: 4; 5

SUMMARY:
The purpose of this study is to define the mechanism(s) through which Obstructive Sleep Apnea/Hypopnea (OSAH) promotes abnormal metabolic processes which characterize the metabolic syndrome. The investigators hypothesize that the sleep fragmentation and intermittent sleep hypoxia which occur in OSAH patients promote oxidative stress and inflammation which in turn lead to insulin resistance, dyslipidemia, abnormal vascular reactivity and other processes which are consistent with the metabolic syndrome.

DETAILED DESCRIPTION:
The metabolic syndrome has been defined as insulin resistance, central obesity, systemic hypertension and dyslipidemia and is associated with increased cardiovascular (CV) risk. Obstructive Sleep Apnea-Hypopnea (OSAH) is also associated with increased CV risk and insulin resistance. Since OSAH is associated with oxidative stress and pro-inflammatory processes, both of which are associated with insulin resistance, it follows that oxidative stress and inflammation may mediate the linkage between OSAH, insulin resistance and ultimately, the metabolic syndrome.

The overall goal of this research is to test the hypothesis that oxidative stress and inflammation link OSAH to insulin resistance as well as other CV risk-promoting conditions reflecting the metabolic syndrome (e.g. hyperlipidemia). We will specifically test if the individual sleep consequences of OSAH, including sleep fragmentation and intermittent sleep hypoxia, promote oxidative stress and inflammation which in turn promote insulin resistance and other features of the metabolic syndrome.

Aim 1a: To determine the effect of sleep fragmentation on oxidative stress and inflammation and features of the metabolic syndrome including insulin resistance, dyslipidemia, obesity, and hypertension.

Aim 1b: To assess the interaction between pre-existing metabolic syndrome and the overweight condition without metabolic syndrome, with regard to the effects of sleep fragmentation on the study variables, we will contrast the effect of experimentally-induced sleep fragmentation in non-OSAH/overweight individuals with the metabolic syndrome, non-OSAH/overweight individuals without metabolic syndrome and a control group of non-OSAH/normal weight without metabolic syndrome.

Aim: 2: To evaluate the effect of intermittent sleep hypoxia on oxidative stress and inflammation and explore the relationships between these two processes and insulin resistance, lipid profile, heart period variability and plasma cortisol.

Aim: 3: Using microarray data from peripheral monocytes, we will explore if specific gene expression patterns after the study conditions are associated with alterations consistent with metabolic syndrome.

Aim: 4: This exploratory aim is to collect preliminary data regarding the correlation among genetic variations (polymorphisms), gene expression patterns (microarray) and resultant protein production (proteomics). These data will be used for hypothesis development.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoker for at least 6 months
* No history of movement disorder during sleep, or circadian rhythm disorder
* No excessive daytime sleepiness
* No history of chronic insomnia, mood or affective disorders or other psychiatric disorders
* Participants maintain a regular sleep-wake pattern with an estimated sleep time between 6.5 and 10 hours per night
* Ability and willingness to avoid meat with its juice (gravy), cured or smoked foods and green leafy vegetables, fruit and fruit juices, food products or vitamin supplements containing vitamin C and E supplements for at least 1 day prior to and during the study periods
* Consumption of less than 1 alcoholic beverage per day
* Ability to understand the study and sign the informed consent
* Not currently pregnant
* Live within 45 miles of the study site
* No uncontrolled hypertension (blood pressure greater than 150/100)
* Willingness to avoid caffeinated beverages and food during the study protocol period

Participants With Sleep Apnea:

* Diagnosis of severe Obstructive Sleep Apnea and Hypopnea (OSAH) (RDI greater than 25) and initiation of positive airway pressure therapy more than 1 month before enrollment
* Must have had an adequate clinical titration of positive airway pressure therapy
* On positive airway pressure for at least 1 month with adherence of more than 5 hours of use per day with no history of snoring, no excessive daytime sleepiness and no reported observed apnea episodes on positive airway pressure
* Willing to sleep with and without positive airway pressure therapy as required by the study protocol

Exclusion Criteria:

* History or physical examination evidence of active coronary artery disease, heart failure, cardiomyopathy, syncope, potentially life-threatening arrhythmia, stroke, transient ischemic attack, neurologic impairment, renal, hepatic or thyroid disease (unless on stable thyroid replacement medication); history of diabetes mellitus; history of cancer within the past 10 years (other than basal cell carcinoma), venous thrombosis, or collagen-vascular disease or other condition that the investigators believe may be exacerbated by participation in the stud
* History of awakening with angina pectoris
* Currently taking medication for mood or affective disorders or that affect heme metabolism, autonomic nervous system or sleep architecture, or prescribed nitrates or corticosteroids
* Physician-diagnosed Alzheimer's or non-Alzheimer's dementia
* Previous surgery for sleep apnea
* Hematocrit less than 32
* Use of a hearing aid in one or both ears
* History of a bleeding disorder, abnormal bleeding, or known adverse reaction to heparin
* Inability to obtain venous blood or a low likelihood of obtaining venous access as required in this protocol
* History of migraine of a nature, frequency, and severity that, in the investigators' judgement, may be precipitated by participation in the protocol
* Presence of a potentially life-threatening dysrhythmia on the clinical diagnostic PSG
* History of motor vehicle accident due to falling asleep; not currently employed as a driver in the transportation industry or an airplane pilot
* Lipid-lowering agents for participants without a history of sleep apnea
* Individuals on positive airway pressure therapy for sleep apnea must not have lost more than 10 pounds of weight since starting this treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2003-09; Primary Completion 2008-08 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
circulating and exhaled biomarkers of oxidative stress and pro-inflammatory cytokines, insulin resistance, lipid profile, plasma cortisol, and heart period variability (a reflection of sympathovagal tone) | before and after 2 consecutive nights

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Sanders, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States